CLINICAL TRIAL: NCT02195089
Title: A Phase 1/2a Trial to Evaluate the Efficacy and the Safety of BLS_ILB_E710c for the Fertile Women With Cervical Intraepithelial Neoplasia(CIN3)
Brief Title: Efficacy and Safety Study of BLS_ILB_E710c for the Fertile Women With Cervical Intraepithelial Neoplasia(CIN3)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioLeaders Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMT2013-BLS-ILB-E710c; 12591 (Other: Ministry of Food and Drug Safety)
Record Dates: First submitted 2014-07-15; First posted 2014-07-21 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Treatment of Cervical Intraepithelial Neoplasia(CIN3)
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BLS_ILB_E710c 500mg (Experimental): * Drug: BLS_ILB_E710c 500mg
  * Dosage and duration: 2 capsules per day for 20 days (week 1,2,4 & 8)
  Interventions: Drug: BLS_ILS_E710c 500mg
- BLS_ILS_E710c 1000mg (Experimental): * Drug: BLS_ILS_E710c 1000mg
  * Dosage and duration: 4 capsules per day for 20 days (week 1,2,4 & 8)
  Interventions: Drug: BLS_ILB_710c 1000mg
- BLS_ILS_E710c 1500mg (Experimental): * Drug: BLS_ILS_E710c 1500mg
  * Dosage and duration: 6 capsules per day for 20 days (week 1,2,4 & 8)
  Interventions: Drug: BLS_ILS_E710c 1500mg

INTERVENTIONS:
Drug: BLS_ILS_E710c 500mg — - 2 capsules per day for 20 days (week 1,2,4 & 8)
  Other Names: CIN3 Theraputic Vaccine
  Arms: BLS_ILB_E710c 500mg
Drug: BLS_ILB_710c 1000mg — - 4 capsules per day for 20 days (week 1,2,4 & 8)
  Other Names: CIN3 Theraputic Vaccine
  Arms: BLS_ILS_E710c 1000mg
Drug: BLS_ILS_E710c 1500mg — - 6 capsules per day for 8 weeks (week 1,2,4 & 8)
  Other Names: CIN3 Theraputic Vaccine
  Arms: BLS_ILS_E710c 1500mg

SUMMARY:
The purpose of this study is to determine the efficacy and the safety of BLS-ILB-E710c for the the fertile women with Cervical Intraepithelial Neoplasia (CIN3).

DETAILED DESCRIPTION:
This study is to see the regression rate of Cervical Intraepithelial Neoplasia (CIN3) and to see the inducement of Cytotoxic T Lymphocyte.

The First treatment group will be administered with BLS-ILB-E710c 500mg for 8 weeks followed by 1 week observation The Second treatment group will be administered with BLS-ILB-E710c 1000mg for 8 weeks followed by 1 week observation The Third treatment group will be administered with BLS-ILB-E710c 1500mg for 8 weeks followed by 1 week observation The fourth treatment group will be administered with BLS-ILB-E710c Optimum dose for 8 weeks followed by 8 weeks observation

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal patients between age of 20 and 50.
* Patients with cervical intraepithelial neoplasia 3(CIN3).
* Only infection with HPV type 16.
* Patients with Capable of observation of all of lesions by Colposcopy biopsy.
* Be informed of the nature of the study and will give written informed consent.
* Be agree with contraception during study
* White Blood Cell Count(WBC) over 4thous/ul, Hemoglobin above over 9.0g/dL Platelet over 150thous/uL and ANC(Absolute Neutrophil Count) over 1,500 /mm^3
* Normal for EKG(Electrocardiography)
* AST/ALT : 2.5 times less than normal range

Exclusion Criteria:

* Autoimmune Disease or Prohibited drug(Therapy) bring about immunosuppressive.
* Patient that has medical history of hypersensitivity about Food containing Lactic acid bacteria or Lactic acid bacteria medication.
* Patient with Acute illness(ex. Acute Appendicitis, Myocardial infarction, Hemorrhage, meningitis etc.)
* Investigational product within three months before the start of the drug administration to patients treated with other test drug.
* Patient with Chronic pancreatitis currently or Patients diagnosed with acute pancreatitis.
* Organopathy Patient with Inflammatory intestine·bowel disease, gastrointestinal tumors, ulcers, bleeding, perforation etc.
* Pregnant or lactating women
* Patient with HBV or HCV infection (except for Asymptomatic)
* Patient that Investigator judge
* Deemed inappropriate for researchers to judge the patient

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2014-03; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Phase 1 : Safety | up to 9 weeks
  Dose Limiting Toxicity(DLT) is assessed by NCI-CTC version 4.0
Phase 2a : Regression rate | screening and 9 weeks(option), 16 weeks.
  Regression rate will be assessed at the time of screening and 9 weeks(option), 16 weeks. Regression means the change from the stage of CIN1 to normal

SECONDARY OUTCOMES:
Reid Colposcopic Index | Phase 1 : up to 9 weeks
  Reid Colposcopic Index will be assessed at the time of screening,4 weeks 9.
Reid Colposcopic Index | Phase 2a : up to 16 weeks
  Reid Colposcopic Index will be assessed at the time of screening,4 weeks, 9 weeks, 12 weeks, 16 weeks
Serum anti-E7 antibody | 1 week, 9 weeks, 16 weeks
  Serum anti-E7 antibody will be assessed at the time of 1 week, 9 weeks, 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Kwan Lee, MD, PhD, Principal Investigator — Korea University Guro Hospital; Tae Jin Kim, MD, PhD, Principal Investigator — Kwandong University College of Medicine Cheil Hospital; Jong Sup Park, MD, PhD, Principal Investigator — The Catholic University, Korea Seoul St Mary's Hospital; Chi-Heum Cho, MD, PhD, Principal Investigator — The Dongsan Medical Center of Keimyung University; Jong Hyeok Kim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (5):
- South Korea (5):
  - Korea University Guro Hospital, Seoul, Seoul
  - The Dongsan Medical Center of Keimyung University, Daegu
  - Kwandong University College of Medicine Cheil Hospital, Seoul
  - The Catholic University, Korea Seoul St Mary's Hospital, Seoul
  - Asan Medical Center, Seoul

REFERENCES:
- [Derived] Park YC, Ouh YT, Sung MH, Park HG, Kim TJ, Cho CH, Park JS, Lee JK. A phase 1/2a, dose-escalation, safety and preliminary efficacy study of oral therapeutic vaccine in subjects with cervical intraepithelial neoplasia 3. J Gynecol Oncol. 2019 Nov;30(6):e88. doi: 10.3802/jgo.2019.30.e88. PMID 31576684